CLINICAL TRIAL: NCT01701661
Title: Compression Therapy Versus Surgery in the Treatment of Superficial Venous Reflux - A Randomized Controlled Trial
Brief Title: Compression Therapy Versus Surgery in the Treatment of Superficial Venous Reflux
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Maarit Venermo, MD,PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TYH4209
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Venous Insufficiency
Keywords: venous surgery; compression therapy
MeSH Terms: conditions — Venous Insufficiency | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conservative treatment (Active Comparator): Compression stockings class II
  Interventions: Other: conservative treatment
- Operative treatment (Active Comparator): stripping of main trunk or if previously removed, removal or ligating the refloating trunk
  Interventions: Procedure: Operative treatment

INTERVENTIONS:
Procedure: Operative treatment — stripping of main trunk or if previously removed, removal or ligating the refluating trunk
  Arms: Operative treatment
Other: conservative treatment — Compression stockings class II
  Arms: conservative treatment

SUMMARY:
Randomized controlled trial, a method used to implement the random allocation sequence is numbered containers.

The aim of the study is to compare compression therapy with compression stockings and surgery eliminating superficial venous reflux in patients with duplex ultrasound verified superficial venous reflux without skin changes or ulceration.

DETAILED DESCRIPTION:
Superficial venous reflux is common in adult population. Uncomplicated disease, where there is no skin changes but varicose veins with or without leg swelling, can be totally asymptomatic but also cause various symptoms as pain, aching and discomfort of leg usually caused by increased venous pressure. Varicose veins may also cause cosmetic problem. Compression stockings relief the symptoms as they normalize venous pressure. In surgical treatment, axial reflux is treated usually by removing incompetent superficial veins. The aim of the study is to compare conservative treatment with compression stockings with surgical treatment of superficial venous reflux. In operative treatment the great saphenous vein or lesser saphenous vein are removed after flush ligation by femoral vein and stripping of the trunk. If the main trunk has been removes previously, axial refluating veins are removed or ligated according to the DUS finding. The patients in both groups are examined at the baseline and followed up to two years by ultrasound scanning. Patients clinical classification, venous disability score, venous disease severity score, anatomical path of reflux as well as quality of life are studied at the baseline, at one year follow-up and two years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic superficial vein insufficiency
* patient must be 20-70 years old
* degree of difficulty of vein insufficiency C2-C3
* venous disability score 1-2
* patient is agreeable to the study

Exclusion Criteria:

* peripheral atherosclerotic occlusive disease
* lymphoedema
* severe concomitant disease (ASA 3-5)
* venous ulcers or unclassified skin changes
* BMI more than 35

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2004-09; Primary Completion 2008-10 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Symptom relief | two years
  Patients are examined at the baseline, one and 2-year follow-up and the following measures are compared: clinical classification, venous disability score, venous disease severity score, reflux according to ultrasound examination.

SECONDARY OUTCOMES:
Quality of life | two years
  Quality of life is evaluated with two questionnaires: Aberdeen (which is a 13-item questionnaire with categories related specially to disadvantages caused by varicose veins) and 15D (a questionnaire with categories related to general quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Maarit Venermo, MD,PhD, Principal Investigator — Department of Vascular Surgery, Helsinki University Central Hospital
Locations (1):
- Department of Vascular Surgery, Helsinki University Central Hospital, Helsinki, HUS, Finland